CLINICAL TRIAL: NCT07228273
Title: A Phase II Randomized Clinical Trial of Venetoclax Combined With FLAG IDA Induction and Consolidation Compared to Standard of Care for Newly Diagnosed Patients With Acute Myeloid Leukemia
Brief Title: Induction and Consolidation With Fludarabine, Cytarabine, Idarubicin, and Venetoclax for the Treatment of Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Curtis Lachowiez, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00028170; NCI-2025-04104 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00028170 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2025-11-12; First posted 2025-11-14 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Specimen Handling; Biopsy; Cytarabine; Daunorubicin; fludarabine; Idarubicin; venetoclax

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (fludarabine, cytarabine, idarubicin, venetoclax) (Experimental): See Detailed Description.
  Interventions: Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Cytarabine; Procedure: Echocardiography Test; Drug: Fludarabine; Drug: Idarubicin; Procedure: Multigated Acquisition Scan; Other: Questionnaire Administration; Drug: Venetoclax
- Arm 2 (cytarabine, daunorubicin) (Active Comparator): INDUCTION: Patients receive cytarabine IV on days 1-7 and daunorubicin IV on days 1-3 of each cycle. Cycles repeat every 28 days for up to 1 cycle in the absence of disease progression or unacceptable toxicity. Patients achieving CR, CRh, CRi, or MLFS after one induction cycle proceed to consolidation. Patients achieving PR after one induction cycle may proceed to consolidation at the investigator's discretion. Patients with ≥ 5% blasts after one induction cycle may receive a second cycle of induction therapy.
  CONSOLIDATION: Participants receive cytarabine IV over 3 hours BID on days 1, 3, and 5 of each cycle. Cycles repeat every 28 days for up to 4 post-induction cycles in the absence of disease progression or unacceptable toxicity.
  Additionally, patients undergo ECHO or MUGA scan during screening and on study as clinically indicated. Patients also undergo bone marrow aspiration and biopsy and blood sample collection throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Cytarabine; Drug: Daunorubicin; Procedure: Echocardiography Test; Procedure: Multigated Acquisition Scan; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
  Arms: Arm 2 (cytarabine, daunorubicin)
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Daunorubicin — Given IV
  Other Names: Daunomycin; Daunorrubicina; DNR; Leukaemomycin C; Rubidomycin; Rubomycin C
  Arms: Arm 2 (cytarabine, daunorubicin)
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
  Arms: Arm 1 (fludarabine, cytarabine, idarubicin, venetoclax)
Drug: Idarubicin — Given IV
  Other Names: 4-Demethoxydaunomycin; 4-Demethoxydaunorubicin; 4-DMDR
  Arms: Arm 1 (fludarabine, cytarabine, idarubicin, venetoclax)
Procedure: Multigated Acquisition Scan — Undergo MUGA scan
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Other: Questionnaire Administration — Ancillary studies
Drug: Venetoclax — Given PO
  Other Names: ABT 199; ABT-0199; ABT-199; ABT199; GDC 0199; GDC-0199; GDC0199; RG7601; Venclexta; Venclyxto
  Arms: Arm 1 (fludarabine, cytarabine, idarubicin, venetoclax)

SUMMARY:
This phase II trial compares induction and consolidation therapy with fludarabine, cytarabine, idarubicin, and venetoclax to cytarabine and daunorubicin induction and cytarabine consolidation for the treatment of acute myeloid leukemia (AML). Patients with AML often receive induction and consolidation therapy. Induction therapy is given first to get the patient's AML under control (remission). Consolidation therapy is given after the cancer has disappeared following the initial therapy. Consolidation therapy is used to kill any cancer cells that may be left in the body. Chemotherapy drugs, such as fludarabine, cytarabine, idarubicin, and daunorubicin, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Venetoclax is in a class of medications called B-cell lymphoma-2 (BCL-2) inhibitors. It may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. Giving fludarabine, cytarabine, idarubicin, and venetoclax for induction and consolidation therapy may be more effective in treating AML.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assess the efficacy of treatment based on rates of measurable residual disease negative composite complete remission (CRc-MRD-) determined using multiparameter flow cytometry (MFC).

SECONDARY OBJECTIVES:

I. Assess the efficacy of treatment based on complete response (CR) disease remission.

II. Assess the efficacy of treatment based on overall clinical response. III. Assess the safety of treatment. IV. Assess survival in the absence of treatment failure, hematologic relapse, or progressive disease.

V. Assess patient survival after commencing study therapy. VI. Assess the delay in hematopoietic stem cell transplant (HSCT) referral and consultation for transition to HSCT.

VII. Assess the efficacy of treatment based on transitioning to HSCT. VIII. Assess disease response after transplant among participants who proceed to HSCT.

IX. Assess risk of post-transplant infection among participants who proceed to HSCT.

X. Assess risk of post-transplant graft versus host disease (GVHD) among participants who proceed to HSCT.

XI. Assess survival in the absence of post-HSCT GVHD and relapse among participants who proceed to HSCT.

EXPLORATORY OBJECTIVES:

I. Evaluate the depth of response with measurable residual disease (MRD) testing and compare methods of determining MRD status.

II. Evaluate survival of measurable residual disease negative (MRD-) patients with CR versus CR with partial or incomplete hematologic recovery.

III. Assess participant quality of life (QoL) using European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ C30).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM 1:

INDUCTION: Patients receive fludarabine intravenously (IV) over 30 minutes and cytarabine IV over 4 hours on days 2, 3, 4, 5, and 6, idarubicin IV over 15-30 minutes on days 4, 5, and 6, and venetoclax orally (PO) once daily (QD) on days 3-9 of each cycle. Cycles repeat every 28 days for up to 1 cycle in the absence of disease progression or unacceptable toxicity. Patients achieving CR, CR with partial hematologic recovery (CRh), CR with incomplete blood count recovery (CRi), or morphologic leukemia-free state (MLFS) after one induction cycle proceed to consolidation. Patients achieving partial response (PR) after one induction cycle may proceed to consolidation at the investigator's discretion. Patients with ≥ 5% blasts after one cycle of induction may receive a second cycle of induction therapy.

CONSOLIDATION: Patients receive fludarabine IV over 30 minutes and cytarabine IV over 4 hours on days 2, 3, and 4 of each cycle, idarubicin IV over 15-30 minutes on days 4, 5, and 6 of either cycles 3 and 6 or cycles 4 and 7, and venetoclax PO QD on days 3-9 of each cycle. Cycles repeat every 28 days for up to 6 post-induction cycles in the absence of disease progression or unacceptable toxicity.

ARM 2:

INDUCTION: Patients receive cytarabine IV on days 1-7 and daunorubicin IV on days 1-3 of each cycle. Cycles repeat every 28 days for up to 1 cycle in the absence of disease progression or unacceptable toxicity. Patients achieving CR, CRh, CRi, or MLFS after one induction cycle proceed to consolidation. Patients achieving PR after one induction cycle may proceed to consolidation at the investigator's discretion. Patients with ≥ 5% blasts after one induction cycle may receive a second cycle of induction therapy.

CONSOLIDATION: Participants receive cytarabine IV over 3 hours twice daily (BID) on days 1, 3, and 5 of each cycle. Cycles repeat every 28 days for up to 4 post-induction cycles in the absence of disease progression or unacceptable toxicity.

Additionally, all patients undergo echocardiography (ECHO) or multigated acquisition (MUGA) scan during screening and on study as clinically indicated. Patients also undergo bone marrow aspiration and biopsy and blood sample collection throughout the trial.

After completion of study treatment, patients are followed up at 30 days and then every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Ability to comprehend the investigational nature of the study and provide written informed consent
* Age 18 to ≤ 65 years (yrs), at the time of consent
* All gender identities, races, or ethnicities are eligible
* Newly documented, previously untreated diagnosis of AML or myelodysplastic syndrome (MDS) with marrow blasts ≥ 10%, in agreement with 2022 European LeukemiaNet criteria (ELN22)

  * Leukapheresis and treatment with cytarabine or hydroxyurea prior to study initiation is permitted for cytoreduction in patients with proliferative disease. NOTE: Treatment with cytarabine is limited to up to 2 grams total at least 14 days prior to starting on protocol defined therapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Willingness to undergo hematopoietic stem cell transplant (HSCT)
* Ability to take medications by mouth or feeding tube
* Adequate hematologic and organ function
* Institutional standards, New York Heart Association (NYHA) criteria for cardiac function
* Calculated creatinine clearance (according to the Cockcroft-Gault equation) > 40 mL/min
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) ≤ 3 x upper limit of normal (ULN), unless considered due to leukemic involvement
* Alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 3 x ULN, unless considered due to leukemic involvement
* Total bilirubin ≤ 1.5 x ULN, unless due to Gilbert's disease or leukemic involvement
* Willing and able to

  * Adhere to study schedule of activities and lifestyle restrictions while on treatment;
  * Provide bone marrow (BM) aspirate and core biopsy samples; AND
  * Accept supportive and prophylactic care for hematologic toxicities, infection, and immediate sequelae, including transfusions
* Negative pregnancy test within 3 days of start of treatment for persons of childbearing potential (PCBP)
* Based on animal studies and the known pharmacology of the study drugs, PCBP and sperm-producing participants who are sexually active with a PCBP must comply with study requirements for contraception

  * PCBP (participants and PCBP partners of participants) must agree to use an approved contraception and to refrain from donating / cryopreserving ova from cycle (C) 1 day (D) 1 until 6 months following the last dose of study treatment
  * Participants who produce viable sperm and who have intercourse with PCBP must agree to use an approved contraception method and to refrain from donating sperm from C1D1 until 3 months following the last dose of study treatment

Exclusion Criteria:

* Documented t(15;17) (acute promyelocytic leukemia [APL]), and/or mutation(s) to FLT3 ITD or core binding factor (CBF). Point mutations within the tyrosine kinase domain (FLT3 TKD) are allowed
* Another active malignancy within the previous 5 years, except treated early stage carcinomas of the skin, or at the investigator's discretion
* Known, active central nervous system (CNS) involvement with AML
* Recent and significant medical interventions, such as major surgery within 28 days of start of treatment
* GVHD or autologous stem cell transplant within 100 days of start of treatment
* Currently receiving investigational therapy or chemotherapy within 28 days, or 5 half-lives, whichever is longer, with the exception of hydroxyurea or cytarabine for cytoreduction purposes
* Prior treatment with a BCL 2 inhibitor within 12 months prior to the start of treatment
* Use of strong or moderate CYP3A4 inducers or inhibitors or P-gp inhibitors within 2 days or 3 half-lives, whichever is longer, prior to start of treatment with venetoclax or at the discretion of the investigator if dose reductions, based on the interaction, have been specified
* History of allergic response to any of the interventional agents or any excipients in the formulations
* Inadequate organ function, including the following (or at the discretion of the investigator):

  * History of New York Heart Association (NYHA) class III or IV congestive heart failure or left ventricular ejection fraction (LVEF) < 40% by echocardiogram (ECHO) or multigated acquisition (MUGA) scan
  * Unstable/uncontrolled angina pectoris, history of severe and/or uncontrolled ventricular arrhythmias, or history of myocardial infarction within the last 6 months
  * A white blood cell count (WBC) > 25 x 10^⁹/L
* Known dysphagia in the absence of a feeding tube, short-gut syndrome, or other conditions or causes that would affect the ingestion and/or gastrointestinal absorption of drugs administered orally
* Active hepatic disorder or documented positive hepatitis B or C virus (HBV/HCV, respectively) status, except in cases of undetectable HBV/HCV viral load for at least 3 months prior to the start of treatment. (Hepatitis B or C testing is not required for eligibility assessment.)
* Individuals with positive serology for human immunodeficiency virus (HIV) who are undergoing treatment with highly active antiretroviral therapy (HAART) (or another therapy that may interfere with metabolism of study agents) are not eligible. If the HIV infection is controlled with another medication type or if an acceptable alternative HIV treatment can be substituted for HAART, enrollment may proceed
* Uncontrolled infection. Participants with controlled infection must be afebrile and hemodynamically stable for at least 72 hours prior to start of treatment and must be amenable to alternate treatment if current treatment will interact with investigational regimen
* Psychiatric illness/social situations that would limit compliance with study requirements
* Unwillingness to stop breastfeeding. Because there is a potential risk for adverse events in nursing infants secondary to treatment of the mother, breastfeeding is not allowed throughout the study for 6 weeks after the last dose of study drug

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-12-12 (Actual); Primary Completion 2029-06-24 (Estimated); Study Completion 2029-08-24 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants achieving measurable residual disease negative composite complete remission (CRc-MRD-) | Up to 30 days post last dose of study drug
  Will be defined as the achievement of both measurable disease negative (MRD-) by multiparameter flow cytometry and complete response (CR), CR with partial hematologic recovery (CRh), or CR with incomplete blood count recovery (CRi). Participants who do not qualify as efficacy-evaluable (usually due to early death or withdrawal because of toxicity) will be considered non-responders. A point estimate and 95% exact confidence interval (CI) for CRc MRD- will be computed for each arm (and time point) separately and the CRc MRD- rate will be statistically compared across arms with Fisher's exact test at 3 timepoints: end of induction, end of the first consolidation cycle, and end of treatment. A Hochberg multiplicity adjustment will be applied to the p-values from these 3 Fisher exact tests to control the family wise error rate (at α=0.05) for between-arm comparisons of the primary endpoint. CRc MRD- status at each of the above-specified time points will be modeled with logistic regression.

SECONDARY OUTCOMES:
Percentage of participants achieving CR | Up to 30 days post last dose of study drug
  Will be computed for each arm separately in both the safety set and the efficacy set. Will be presented with a point estimate and exact binomial 95% CI. will also be modeled with logistic regression with baseline patient and disease features as predictors and results considered hypothesis-generating.
Percentage of participants achieving composite complete remission (CRc) | Up to 30 days post last dose of study drug
  CRc will be defined as the achievement of CR, CRh, or CRi. Will be computed for each arm separately in both the safety set and the efficacy set. Will be presented with a point estimate and exact binomial 95% CI. will also be modeled with logistic regression with baseline patient and disease features as predictors and results considered hypothesis-generating.
Percentage of participants achieving an overall response (ORR) | Up to 30 days post last dose of study drug
  Will be defined as the proportion of participants who attain a partial remission (PR) or better (i.e., CR, CRh, CRi, morphologic leukemia-free state, or PR) after receiving study treatment. Will be computed for each arm separately in both the safety set and the efficacy set and presented with point estimate and exact binomial 95% CI. Will also be modeled with logistic regression with baseline patient and disease features as predictors and results considered hypothesis-generating.
Incidence of treatment-emergent grade ≥ 3 adverse events (AEs) | Up to 30 days after the last dose of any study drug
  Will be assessed using Common Terminology Criteria for Adverse Events version 5.0. The incidence of specific grade ≥ 3 AEs will be reported with frequencies and percentages, at the overall participant level and by grade, attribution (i.e., a separate table for treatment-related AEs), and seriousness (i.e., separate tables for serious adverse events).
Event free survival (EFS) | From cycle (C)1 day(D)1 to first occurrence of treatment failure, disease progression, or death due to any cause, assessed up to 2 years
  If these events do not occur prior to end of study (EOS), participant is censored at date of last disease assessment. Will be estimated for the efficacy set using the Kaplan-Meier method, with median EFS and EFS rates at common landmark times (e.g., 6 months, 1 year, 2 years) presented with 95% log-log CIs. Cox models will be fit to EFS to assess the impact of baseline patient and disease features, with model results (i.e., hazard ratios and Wald test p-values) interpreted as hypothesis-generating.
Overall survival (OS) | From C1D1 to date of death due to any cause, assessed up to 2 years
  If no death occurs prior to EOS, participant is censored at last known alive date. Will be computed in each arm for both the safety set and the efficacy set. Will be estimated with the Kaplan-Meier method. Median OS and OS rates at common landmark times (e.g., 1 year, 2 years) will be estimated with 95% log-log CIs. For each of the two specified analysis sets, Cox models will be fit to OS to assess the impact of baseline patient and disease features and hematopoietic stem cell transplant (HSCT) as a time-dependent covariate, with results considered hypothesis generating.
Time to HSCT referral | Up to 2 years after end of study treatment
  Within each arm and for both the safety and efficacy sets (separately), cumulative incidence functions (CIFs) will be used to estimate the post-C1D1 time to HSCT referral with death considered a competing risk and patients lacking these bone marrow transplant (BMT) preparation related events being censored at EOS. Between arm differences in time to each of these HSCT-preparatory events will be computed using Gray's test. For each participant cohort (i.e., within each arm for both the safety and efficacy sets), the proportion of patients who are referred to HSCT will be computed with point estimate and 95% exact binominal CI. Fisher's exact test will be employed to test for an association between the occurrence of each HSCT-preparatory event and study arm.
Time to completed consult for HSCT | Up to 2 years after end of study treatment
  Within each arm and for both the safety and efficacy sets (separately), CIFs will be used to estimate the post-C1D1 time to HSCT consultation with death considered a competing risk and patients lacking these BMT preparation related events being censored at EOS. Between arm differences in time to each of these HSCT-preparatory events will be computed using Gray's test. For each participant cohort (i.e., within each arm for both the safety and efficacy sets), the proportion of patients who complete a HSCT consult will be computed with point estimate and 95% exact binominal CI. Fisher's exact test will be employed to test for an association between the occurrence of each HSCT-preparatory event and study arm.
Percentage of participants who transition to HSCT | Up to 2 years after end of study treatment
  Will be computed on both the safety and efficacy sets within each study arm. Besides a point estimate and exact binominal 95% CI for the proportion of patients proceeding to HSCT at any time or within 100 days of commencing study therapy, time-to-HSCT (measured from C1D1) will be estimated within each arm using a CIF, tested across arms with Gray's test, and modeled with Fine-Gray regressions (with baseline patient and disease features as predictors and results considered as hypothesis-generating). For these analyses, pre-HSCT deaths will be considered a competing risk and patients alive but not transplanted will be censored when going off-study.
Cumulative incidence of HSCT | Up to 2 years after end of study treatment
  Will be computed on both the safety and efficacy sets within each study arm. Besides a point estimate and exact binominal 95% CI for the proportion of patients proceeding to HSCT at any time or within 100 days of commencing study therapy, time-to-HSCT (measured from C1D1) will be estimated within each arm using a CIF, tested across arms with Gray's test, and modeled with Fine-Gray regressions (with baseline patient and disease features as predictors and results considered as hypothesis-generating). For these analyses, pre-HSCT deaths will be considered a competing risk and patients alive but not transplanted will be censored when going off-study.
Percentage of participants who are MRD- post-HSCT | From HSCT day 0 to day +365 post-HSCT
  Will be estimated along with an exact binomial 95% CI.
Cumulative incidence of grade 2-3 post-HSCT infections | From HSCT day 0 to day +100 post-HSCT
  Will be assess moderate and severe bacterial, viral, and fungal infections according to Blood and Marrow Transplant Clinical Trials Network criteria. Will be estimated with a CIF (considering death as a competing risk).
Cumulative incidence of grade ≥ II acute graft versus host disease (aGVHD) | From HSCT day 0 to day +365 post-HSCT
  Will be assessed using the Mount Sinai Acute Graft Versus Host Disease International Consortium (MAGIC) criteria. Will be estimated with a CIF (considering death as a competing risk).
Cumulative incidence of grade ≥ 2 chronic graft versus host disease (cGVHD) | From HSCT day 0 to day +365 post-HSCT
  Will be assessed using the National Institutes of Health consensus criteria. Will be estimated with a CIF (considering death as a competing risk).
GVHD-free, relapse-free survival (GRFS) | From HSCT day 0 to disease relapse, MAGIC grade III-IV aGVHD, cGVHD requiring systemic therapy, death from any cause or last known alive, or day + 365 post-HSCT, whichever occurs earliest
  Will be computed and reported for the transplanted population from the time of transplant to a qualifying event. Data from participants without any of the specified GRFS events will be censored at the date of the last disease assessment or the date of the last GVHD assessment, whichever occurs earlier. GRFS will be presented with a point estimate and exact binomial CI.

CONTACTS AND LOCATIONS:
Overall Officials: Curtis A Lachowiez, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States